CLINICAL TRIAL: NCT05463614
Title: Population Pharmacokinetics of Propafenone and Propranolol in Children Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Wei Zhao, professor, Shandong University
Other Study IDs: 2021_Cardiology Drugs_001
Record Dates: First submitted 2022-07-08; First posted 2022-07-19 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Arrhythmia
MeSH Terms: conditions — Arrhythmias, Cardiac | interventions — Propafenone; Propranolol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Propafenone and Propranolol — Propafenone Hydrochloride Tablets, 100-200mg, 1 or 2 times per day; Propranolol Hydrochloride Sustained-Release Capsules, 40mg, 1 times per day

SUMMARY:
The use of propafenone and propranolol in children during clinical treatment was depending mostly on experience. Besides, there was no recommended dose for children in drug instruction. Therefore, the investigators' aim is to study the pharmacokinetics and pharmacodynamics in children.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≤18years. Parental written consent to participate in the study. Patients treat with Propafenone and Propranolol

Exclusion Criteria:

* Patients can not complete the research; Abnormal hepatic and renal function; Patient is allergic to propafenone; There are conditions that researchers do not consider it appropriate to join the research.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: children aged 0-18 years and receive treatment with Propafenone and Propranolol
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Ventricular premature beats of 24 hours | From date of randomization until the date of discharge, assessed up to 12 months
  frequency of Ventricular premature beats of 24 hours

SECONDARY OUTCOMES:
P-R interval | From date of randomization until the date of discharge, assessed up to 12 months
  P-R interval time
QT interval | From date of randomization until the date of discharge, assessed up to 12 months
  QT interval time

CONTACTS AND LOCATIONS:
Locations (1):
- Hebei province Children's Hospital, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: No